CLINICAL TRIAL: NCT03616821
Title: A 54-Week, Multicenter, Randomized, Double-blind, Placebo Controlled, Parallel-group Phase 2 Study to Assess the Efficacy and Safety of Brazikumab in Participants With Moderately to Severely Active Ulcerative Colitis (Expedition Lead-in)
Brief Title: Placebo-Controlled Study of Brazikumab in Participants With Moderately to Severely Active Ulcerative Colitis
Acronym: Expedition
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic decision to discontinue the development of brazikumab in inflammatory bowel disease.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5272C00001; Legacy #3151-201-008 (Other: Allergan); 2018-001605-93 (EudraCT Number); NCT04718818 (obsolete NCT alias)
Record Dates: First submitted 2018-08-01; First posted 2018-08-06 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-10

CONDITIONS: Ulcerative Colitis; IBD
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: Global, multicenter, randomized, double-blind, placebo-controlled, parallel-group, Phase 2 study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Brazikumab Dose 1 (Experimental): Intravenous brazikumab on day 1, day 15, and day 43 followed by Subcutaneous brazikumab every 4 weeks beginning on day 71 through week 50
  Interventions: Drug: Brazikumab
- Brazikumab Dose 2 (Experimental): Intravenous brazikumab on day 1, day 15, and day 43 followed by Subcutaneous brazikumab every 4 weeks beginning on day 71 through Week 50
  Interventions: Drug: Brazikumab
- Placebo (Placebo Comparator): Intravenous placebo on day 1, day 15, and day 43 followed by Subcutaneous every 4 weeks beginning on day 71 through Week 50.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Brazikumab — Intravenous brazikumab on day 1, day 15, and day 43 followed by Subcutaneous brazikumab every 4 weeks beginning on day 71 through Week 50
  Arms: Brazikumab Dose 1; Brazikumab Dose 2
Drug: Placebo — Intravenous placebo on day 1, day 15, and day 43 followed by Subcutaneous placebo every 4 weeks beginning on Day 71 through Week 50.
  Arms: Placebo

SUMMARY:
The present study (D5272C00001/Legacy #3151-201-008) aims to evaluate the efficacy and safety of brazikumab in patients with moderately to severely active UC and will include assessments of clinical responses as demonstrated by improvement of symptoms and of colonic mucosal appearance as observed on endoscopy

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent
2. Aged 18 to 80 years of age
3. Diagnosis of UC with an onset of symptoms for a minimum of 3 months prior to Screening
4. Evidence of UC extending proximal to the rectum (≥ 15 cm of involved colon)
5. Moderately to severely active UC as defined by:

   1. Average daily mMS Stool Frequency subscore ≥ 1 AND Average daily mMS Rectal Bleeding subscore ≥ 1
   2. Modified Mayo endoscopic subscore of ≥ 2 based on a full colonoscopy within 14 days prior to randomization.
6. Participant had an inadequate response or intolerance to intervention with conventional treatment or prior biological treatment or demonstrated CS dependence for the treatment of UC. For participants who have previously used biological treatment, a participant may have failed up to 3 biologics that include up to 2 different mechanisms of action.
7. Participants taking 5-aminosalicylates, oral prednisone (or equivalent), oral budesonide, or immunomodulators must be at a stable dose or discontinued. Topical (rectal) aminosalicylic acid or topical (rectal) steroids should be discontinued.
8. Female participants of childbearing potential must have a negative urine pregnancy test prior to administration of study intervention and must agree to use a highly effective method of birth control throughout the study and for at least 18 weeks after the last dose of study intervention.
9. Women not of childbearing potential are defined as women who are either permanently sterilized (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), or who are postmenopausal.
10. Non sterilized males who are sexually active with a female partner of childbearing potential should use condoms during treatment and until the end of relevant systemic exposure in the male participant, plus a further 18 weeks.
11. No known history of active TB or latent TB without completion of appropriate intervention and negative QFT-TB during Screening.

Complete inclusion criteria are in the Clinical Study Protocol

Exclusion Criteria:

1. Participant has UC limited to the rectum (ie, not beyond 15 cm of the anal verge).
2. Current diagnosis of fulminant colitis, a diagnosis of CD or indeterminate colitis, presence or history of a fistula consistent with CD, primary sclerosing cholangitis, celiac disease, or untreated bile acid malabsorption. Participants with a history of toxic megacolon within 12 months of screening are excluded.
3. History of subtotal colectomy with ileorectostomy or colectomy with ileoanal pouch, Koch pouch, ileostomy, or other prior colonic resection, or need for surgical intervention for control of UC anticipated within 6 months.
4. Participant has received the following treatment:

   1. Infliximab: within 8 weeks prior to randomization.
   2. Adalimumab, certolizumab pegol, or golimumab: within 8 weeks prior to randomization.
   3. Vedolizumab or ustekinumab within 12 weeks of randomization.
   4. Other prohibited medication, biologic or small molecule treatment within 5 half-lives prior to randomization.
   5. Fecal microbiota transplantation: within 8 weeks prior to randomization.
5. Criterion deleted as part of Amendment 5 v6.0
6. Except for ustekinumab, prior exposure to any biologic agent targeting IL-12 or IL-23.
7. Known history of allergy to the study intervention formulation or any of its excipients or components of the delivery device, or to any other biologic therapy.
8. Participant received cyclosporine, mycophenolate mofetil, sirolimus (rapamycin), thalidomide, tacrolimus (FK-506), or tofacitinib within 2 weeks prior to Screening.
9. Participants who received IV or intramuscular steroids within 2 weeks prior to Screening.
10. Participant is currently enrolled in another investigational device or drug study, or is within 35 days or 5 half-lives, whichever is longer, since ending another investigational device or drug study(s), or receiving other investigational agent(s).
11. Participant received a transfusion of blood, plasma, or platelets within 30 days prior to Screening.
12. Participant received a Bacille Calmette-Guérin vaccination within 12 months of randomization or any other live vaccine less than 4 weeks prior to randomization.
13. Participant has any of the following criteria related to infections:

    1. Evidence of a recent systemic fungal infection, requiring inpatient hospitalization, and/or antifungal treatment.
    2. Any infection requiring hospitalization or treatment with IV anti-infectives within 4 weeks of Screening.
    3. Cytomegalovirus or Epstein-Barr virus infection that has not resolved within 8 weeks prior to Screening.
    4. Clinically significant chronic infection that has not resolved within 8 weeks of Screening.
    5. Nonserious infection requiring oral anti-infectives within 2 weeks prior to randomization must be further discussed with study medical monitor.
    6. Clinical evidence of or suspected to have an abscess during Screening.
    7. Any underlying condition that predisposes the participant to infections.
    8. Participant had previous allogenic bone marrow transplant or history of organ or cell-based transplantation.
    9. Clinically significant active infection or signs/symptoms of infection that has the potential to worsen with immunosuppressive therapy.
    10. Signs or symptoms of ongoing infection due to intestinal pathogens.
14. Participant has known or suspected history of chronic use of NSAIDs and/or opiates, drug, or alcohol abuse.
15. History of cancer with the following exceptions: history of basal cell carcinoma and/or squamous cell carcinoma of the skin OR carcinoma in situ of the cervix; with apparent successful curative therapy, greater than 12 months prior to Screening.
16. Clinically significant cardiovascular conditions.
17. Prolonged QTcF interval or conditions leading to additional risk for QT prolongation.
18. Clinically significant kidney disease
19. Abnormal laboratory results at Screening as defined in the study protocol
20. Participant is pregnant or breastfeeding or plans to become pregnant during the study.
21. Participant has other known, pre-existing, clinically significant medical conditions that are not associated with UC and are uncontrolled with standard treatment.
22. Participant has any disorder that may compromise the ability of the participant to give written informed consent and/or to comply with all required study procedures.
23. Employees of the clinical study site or any other individuals involved with the conduct of the study, or immediate family members of such individuals.

Complete exclusion criteria are in the Clinical Study Protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with clinical remission | at Week 10
  Clinical remission defined as: Modified Mayo Score (mMS): Endoscopy subscore = 0 or 1, AND Rectal bleeding subscore = 0, AND Stool frequency subscore = 0 or 1 AND at least a 1 point decrease from baseline

SECONDARY OUTCOMES:
Percentage of participants with sustained clinical remission | at both Week 10 and Week 54
  Sustained clinical remission defined as Modified Mayo Score (mMS): Endoscopy subscore = 0 or 1, AND Rectal bleeding subscore = 0, AND Stool frequency subscore = 0 or 1 AND at least a 1 point decrease from baseline
Percentage of participants with CS-free clinical remission | at Week 54 for patients who are CS-free for at least the last 12 weeks before the assessment at Week 54
  CS-free clinical remission defined as mMS: Endoscopy subscore = 0 or 1, AND Rectal bleeding subscore = 0, AND Stool frequency subscore = 0 or 1 AND at least a 1 point decrease from baseline
Percentage of participants with clinical response | at Week 10
  Clinical response is defined as Reduction in mMS ≥ 2 points from baseline AND ≥ 30% from baseline AND a decrease in the rectal bleeding score ≥ 1 point from baseline or a score of 0 or 1
Percentage of participants with endoscopic improvement | at Week 10
  Endoscopic improvement is defined as Endoscopy subscore ≤ 1
Serum concentration of brazikumab | through Week 68
  Pharmacokinetics: concentration of brazikumab in serum
For each dose level: LS mean of Mayo score and brazikumab pre-dose blood concentration | at 12 weeks after dosing
  Exposure-response
Incidence of anti-drug antibodies | through week 68
  Immunogenicity: incidence of brazikumab anti-drug antibodies in serum
Number and percentage of participants with adverse events | through Week 68
  Number and percentage of patients with reported adverse events.
Percentage of participants with potentially clinically significant changes in laboratory values | through Week 68
  Percentage of patients with potentially clinically significant changes in hematology, clinical chemistry, urinalysis.
Percentage of participants with potentially clinically significant changes in vital signs | through Week 68
  Percentage of patients with potentially clinically significant changes in systolic and diastolic blood pressure, and pulse rate.
Clinically relevant abnormal findings at physical exam | through Week 68
  New or aggregated clinical relevant abnormal medical finding are reported as AE unless related to the disease under study
Percentage of participants with potentially clinically significant changes in ECGs | through Week 68
  Percentage of patients with potentially clinically significant changes in 12-lead ECG recordings

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Bohannon, Study Director — AstraZeneca
Locations (115):
- United States (45):
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Chula Vista, California
  - Research Site, Lancaster, California
  - Research Site, Lincoln, California
  - Research Site, Mission Hills, California
  - Research Site, Poway, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Clearwater, Florida
  - Research Site, Inverness, Florida
  - Research Site, Kissimmee, Florida
  - Research Site, Lakeland, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Naples, Florida
  - Research Site, New Port Richey, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Gurnee, Illinois
  - Research Site, Oak Lawn, Illinois
  - Research Site, Brownsburg, Indiana
  - Research Site, Evansville, Indiana
  - Research Site, Shawnee Mission, Kansas
  - Research Site, Topeka, Kansas
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Marrero, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Wyoming, Michigan
  - Research Site, Biloxi, Mississippi
  - Research Site, Las Vegas, Nevada
  - Research Site, New York, New York
  - Research Site, Sunnyside, New York
  - Research Site, Morehead City, North Carolina
  - Research Site, Beachwood, Ohio
  - Research Site, Springfield, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Uniontown, Pennsylvania
  - Research Site, Amarillo, Texas
  - Research Site, Carrollton, Texas
  - Research Site, Houston, Texas
  - Research Site, Humble, Texas
  - Research Site, Pflugerville, Texas
  - Research Site, San Antonio, Texas
  - Research Site, North Chesterfield, Virginia
- Research Site, Chicoutimi, Quebec, Canada
- Czechia (4):
  - Research Site, Brno
  - Research Site, České Budějovice
  - Research Site, Hradec Králové
  - Research Site, Ostrava
- Germany (3):
  - Research Site, Hamburg
  - Research Site, Kiel
  - Research Site, Ulm
- Research Site, Debrecen, Hungary
- India (6):
  - Research Site, Bangalore
  - Research Site, Hyderabad
  - Research Site, Jaipur
  - Research Site, New Delhi
  - Research Site, Rajkot
  - Research Site, Surat
- Israel (3):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Petah Tikva
- Italy (4):
  - Research Site, Milan
  - Research Site, Negrar
  - Research Site, Rho
  - Research Site, Roma
- Japan (14):
  - Research Site, Asahikawa-shi
  - Research Site, Chiba
  - Research Site, Fukuoka
  - Research Site, Fukuyama-shi
  - Research Site, Hakodate-shi
  - Research Site, Kasama-shi
  - Research Site, Kashiwa-shi
  - Research Site, Koshigaya-shi
  - Research Site, Kure-shi
  - Research Site, Minatoku
  - Research Site, Nagaoka-shi
  - Research Site, Onga-gun
  - Research Site, Sapporo
  - Research Site, Takarazuka-shi
- Poland (13):
  - Research Site, Bydgoszcz
  - Research Site, Chojnice
  - Research Site, Częstochowa
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Ksawerów
  - Research Site, Piaseczno
  - Research Site, Poznan
  - Research Site, Rzeszów
  - Research Site, Sopot
  - Research Site, Torun
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Research Site, San Juan, Puerto Rico
- Russia (6):
  - Research Site, Aramil
  - Research Site, Izhevsk
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Perm
  - Research Site, Tomsk
- Research Site, Košice, Slovakia
- South Africa (3):
  - Research Site, Bloemfontein
  - Research Site, Cape Town
  - Research Site, Plumstead
- South Korea (4):
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Seoul
  - Research Site, Wŏnju
- Research Site, Valencia, Spain
- Taiwan (2):
  - Research Site, Taichung
  - Research Site, Taipei
- Ukraine (2):
  - Research Site, Kyiv
  - Research Site, Vinnytsia
- Research Site, West Bromwich, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home